CLINICAL TRIAL: NCT02296684
Title: Immunotherapy With MK-3475 in Locoregionally Advanced, Surgically Resectable Head and Neck Squamous Cell Carcinoma
Brief Title: Immunotherapy With MK-3475 in Surgically Resectable Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201412118
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Results first posted 2023-05-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Cancer of Head and Neck; Head and Neck Cancer; Neoplasms, Head and Neck; Carcinoma, Squamous Cell of Head and Neck; Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma, Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Neoadjuvant Therapy; Surgical Procedures, Operative; Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided; Cisplatin; Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 (Experimental): * MK-3475 will be given intravenously once approximately 2-3 weeks prior to standard of care surgery.
  * Adjuvant therapy will be dictated by surgical pathology and occurs after standard of care surgery and will consist of:
    * risk-based intensity modulated radiation therapy consisting of 60 Gy in 2 Gy once-daily fraction size (total of 30 fractions)once-daily fraction size (total of 30 fractions)
    * optional image-guided radiation therapy
    * risk-based cisplatin administered intravenously on Days 1, 22, and 43 of treatment course
    * MK-3475 will be given intravenously once every 3 weeks for a maximum of 6 doses if participant is considered high-risk based surgical pathology from standard of care surgery. These doses of MK-3475 will be given after surgery and after all acute toxicities of post-operative standard of care chemotherapy and radiation have resolved to grade 1 or less.
  Interventions: Biological: MK-3475 (neoadjuvant); Procedure: Surgery; Radiation: Intensity modulated radiation therapy; Radiation: Image-guided radiation therapy; Drug: Cisplatin; Biological: MK-3475 (adjuvant); Procedure: Peripheral blood
- Cohort 2: Neoadjuvant MK-3475 (Experimental): -MK-3475 will be given once intravenously and then given again 21 days after dose 1 (14-24 days before standard of care surgery)
  Interventions: Biological: MK-3475 (neoadjuvant); Procedure: Surgery; Radiation: Intensity modulated radiation therapy; Radiation: Image-guided radiation therapy; Drug: Cisplatin; Procedure: Peripheral blood

INTERVENTIONS:
Biological: MK-3475 (neoadjuvant)
  Other Names: SCH 900475; Pembrolizumab; Keytruda
Procedure: Surgery — Standard of care
Radiation: Intensity modulated radiation therapy — Recommended, standard of care
  Other Names: IMRT
Radiation: Image-guided radiation therapy — Recommended, standard of care
  Other Names: IGRT
Drug: Cisplatin — Standard of care
  Other Names: cis-DDP; cis-Platinum II; cis-Diamminedichloroplatinum; DDP
Biological: MK-3475 (adjuvant)
  Other Names: SCH 900475; Pembrolizumab; Keytruda
  Arms: Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475
Procedure: Peripheral blood — -Baseline, time of surgery (between day 14-24 inclusive), 3 months post surgery, 6 months post surgery, 9 months post surgery, 12 months post surgery

SUMMARY:
The goal of this trial is to test the ability of MK-3475 (pembrolizumab) to improve locoregional recurrence and distant metastatic rates in high-risk patients with locally advanced head and neck squamous cell carcinomas (HNSCCs) that are treated with current standard of care surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage III or IV HNSCC oral cavity, hypopharynx, oropharynx, larynx (excluding p16 or HPV-positive oropharynx primaries and sinonasal primaries).
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam by RECIST 1.1.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 x IULN OR Direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (or ≤ 5 x IULN for patients with liver metastases)
  * Serum creatinine ≤ 1.5 x IULN OR Creatinine clearance by Cockcroft-Gault ≥ 30 mL/min/1.73 m2 for patients with creatinine levels > 1.5 x IULN
  * INR ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
* Sexually active women of childbearing potential and men must agree to use 2 methods of contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 120 days after last dose of MK-3475. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment for head and neck cancer.
* Patients with HPV-positive or p16-positive oropharyngeal SCCA.
* Patients with sinonasal SCCAs
* Patients with metastatic SCCA neck disease with an unknown primary tumor site
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Received a live vaccine within 30 days prior to the first dose of MK-3475. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated viruses and are not allowed.
* A history of other malignancy ≤ 3 years previous with the exception of previous head and neck cancer treated only by surgery, basal cell or squamous cell carcinoma of the skin which were treated with local resection only, or carcinoma in situ of the cervix.

Note: patients with synchronous head and neck cancer primaries are an exception to this criterion and may qualify for the study.

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of MK-3475.
* Currently receiving any other investigational agents or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of MK-3475.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, immunosuppression, autoimmune conditions, underlying pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Pregnant and/or breastfeeding. Patient must have a negative serum or urine pregnancy test within 72 hours of study entry.
* Known history of active TB (bacillus tuberculosis).
* Known history of hepatitis B (defined as hepatitis B survace antigen [HBsAg] reactive) or known active hepatitis C (defined as HCV RNA [qualitative] is detected) infection. Note: know testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
* Known history of HIV (HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2025-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uppaluri R, Campbell KM, Egloff AM, Zolkind P, Skidmore ZL, Nussenbaum B, Paniello RC, Rich JT, Jackson R, Pipkorn P, Michel LS, Ley J, Oppelt P, Dunn GP, Barnell EK, Spies NC, Lin T, Li T, Mulder DT, Hanna Y, Cirlan I, Pugh TJ, Mudianto T, Riley R, Zhou L, Jo VY, Stachler MD, Hanna GJ, Kass J, Haddad R, Schoenfeld JD, Gjini E, Lako A, Thorstad W, Gay HA, Daly M, Rodig SJ, Hagemann IS, Kallogjeri D, Piccirillo JF, Chernock RD, Griffith M, Griffith OL, Adkins DR. Neoadjuvant and Adjuvant Pembrolizumab in Resectable Locally Advanced, Human Papillomavirus-Unrelated Head and Neck Cancer: A Multicenter, Phase II Trial. Clin Cancer Res. 2020 Oct 1;26(19):5140-5152. doi: 10.1158/1078-0432.CCR-20-1695. Epub 2020 Jul 14. PMID 32665297
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Assigned to an Arm (Cohort): -Participants who did not receive any treatment and were not assigned to an arm (cohort).
Period: Overall Study
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475 | Not Assigned to an Arm (Cohort)
Started | 36 | 30 | 1
Completed | 34 | 29 | 0
Not Completed | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475 | Not Assigned to an Arm (Cohort) | Total
Number analyzed (Participants) | 36 | 30 | 1 | 67
Age, Continuous [Median (Full Range); unit: years] | 59.5 [32 to 87] | 62.5 [29 to 82] | 51 [51 to 51] | 61 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 0 | 20
  Male | 26 | 20 | 1 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 34 | 29 | 1 | 64
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 0 | 8
  White | 29 | 28 | 0 | 57
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 30 | 1 | 67

OUTCOME MEASURES:

1. Primary Outcome: Locoregional Recurrence Rates in Cohorts 1 and 2
Description: -The percentage of participants who developed local-regional recurrence within one year of surgery
Time Frame: Within 1 year of surgery (surgery occurred within 13-22 days after neoadjuvant MK-3475 dose)
Population: Evaluable Cohort 1 participants for this outcome measure were those who had a high-risk pathology in the surgical specimen after one dose of neoadjuvant MK-3475 (pembrolizumab).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Neoadjuvant MK-3475: -MK-3475 will be given once intravenously and then given again 21 days after dose 1 (14-24 days before standard of care surgery
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
Number analyzed (Participants) | 18 | 30
Participants | 2 | 2

2. Primary Outcome: Distant Failure Rate in Cohorts 1 and 2
Description: -The percentage of participants who developed distant failure within one year of surgery. Distant disease is cancer that is found in another part of the body that is far away from where the original (primary) tumor first formed.
Time Frame: Within 1 year of surgery (surgery occurred within 13-22 days after neoadjuvant MK-3475 dose)
Population: -Evaluable Cohort 1 participants for this outcome measure were those who had a high-risk pathology in the surgical specimen after one dose of neoadjuvant MK-3475 (pembrolizumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
Number analyzed (Participants) | 18 | 30
Participants | 3 | 1

3. Primary Outcome: Rate of Major Pathologic Treatment Effect in Cohort 1
Description: * Major pathologic treatment effect=pathologic tumor response (pTR).
  * pTR was defined as the presence of tumor cell necrosis and keratinous debris with giant cell/histiocytic reaction, quantified as a percentage of the overall tumor bed (area pathologic response/area pathologic response plus viable tumor): pTR-0 (>10%), pTR-1 (10-49%), and pTR-2 (≥50%).
Time Frame: At the time of surgery (surgery occurred within 13-22 days after neoadjuvant MK-3475 dose)
Population: Only those participants enrolled in Cohort 1 were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
Number analyzed (Participants) | 36 | 0
Participants
  pTR-0 | 20 |
  pTR-1 | 8 |
  pTR-2 | 8 |

4. Primary Outcome: Rate of Major Pathologic Treatment Effect in Cohort 2
Description: as for outcome 3
Time Frame: At the time of surgery (surgery occurred within 13-22 days after last neoadjuvant MK-3475 dose)
Population: Only those participants enrolled in Cohort 2 were evaluable for this outcome measure. One participant in Cohort 2 not evaluable for this outcome measure because the participant did not have surgery. One participant in Cohort 2 not evaluable because the data was missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
Number analyzed (Participants) | 0 | 28
Participants
  pTR-0 |  | 13
  pTR-1 |  | 2
  pTR-2 |  | 13

5. Secondary Outcome: Number of Participants in Cohort 1 and 2 Who Experienced Reportable Adverse Events
Description: Reportable adverse events will be tracked for 30 days following the last day of study treatment. For the purposes of this protocol, reportable adverse events are events thought to be possibly, probably, or definitely related to MK-3475. Events thought to be probably or definitely related to surgery, adjuvant chemotherapy, or radiotherapy need not be recorded.
Time Frame: Through 30 days after last dose of MK-3475
Population: Only 12 participants in Cohort 1 received adjuvant MK-3475.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
Number analyzed (Participants) | 36 | 30
Participants
  Grades 1-2 fatigue (neoadjuvant period) | 2 | 3
  Grades 1-2 fever (neoadjuvant period) | 1 | 0
  Grades 1-2 tumor flare (neoadjuvant period) | 1 | 0
  Grades 1-2 AST increase (neoadjuvant period) | 0 | 2
  Grades 1-2 ALT increase (neoadjuvant period) | 0 | 2
  Grades 1-2 fatigue (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 1-2 fatigue (adjuvant period) | 2 | 0
  Grades 1-2 hypothyroidism (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 1-2 hypothyroidism (adjuvant period) | 3 | 0
  Grades 3-4 hypothyroidism (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 3-4 hypothyroidism (adjuvant period) | 1 | 0
  Grades 1-2 AST increase (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 1-2 AST increase (adjuvant period) | 1 | 0
  Grades 1-2 ALT increase (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 1-2 ALT increase (adjuvant period) | 1 | 0
  Grades 1-2 alkaline phosphatase increase (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 1-2 alkaline phosphatase increase (adjuvant period) | 1 | 0
  Grades 1-2 diarrhea (adjuvant period): number analyzed (Participants) | 12 | 0
  Grades 1-2 diarrhea (adjuvant period) | 1 | 0

6. Secondary Outcome: Number of Surgical Complications and/or Delays in Cohorts 1 and 2
Time Frame: At the time of surgery (approximately 2-3 weeks after registration)
Population: One participant in Cohort 2 is not evaluable for the outcome measure because the participant did not have surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
Number analyzed (Participants) | 36 | 29
Participants | 5 | 6

7. Secondary Outcome: Locoregional Recurrence Rates in Cohorts 1 and 2
Time Frame: Through completion of follow-up (estimated to be 5 years after treatment)
Reporting Status: Not Posted

8. Secondary Outcome: Rate of Distant Metastases (DM) in Cohorts 1 and 2
Time Frame: Through completion of follow-up (estimated to be 5 years after treatment)
Reporting Status: Not Posted

9. Secondary Outcome: Event-free Survival (EFS) in Cohorts 1 and 2
Description: Event-free survival will be defined as time from surgery to time to disease recurrence, distant metastasis, new primary, or death due to any cause, whichever occurred first.
Time Frame: Through completion of follow-up (estimated to be 5 years after treatment)
Reporting Status: Not Posted

10. Secondary Outcome: Event-free Survival (EFS) Rate Differences by Presence Versus Absence of Recurrent Genomic Alterations in Cohorts 1 and 2
Description: as for outcome 9
Time Frame: Through completion of follow-up (estimated to be 5 years after treatment)
Reporting Status: Not Posted

11. Secondary Outcome: Overall Survival (OS) Rates Differences by Presence Versus Absence of Recurrent Genomic Alterations in Cohorts 1 and 2
Description: Overall survival will be defined as time from surgery to death from any cause.
Time Frame: Through completion of follow-up (estimated to be 5 years after treatment)]
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For patients who did not receive adjuvant MK-3475 (pembrolizumab), adverse events were tracked for 30 days following the date of surgery. For patients who received adjuvant MK-3475 (pembrolizumab), adverse events were tracked for 30 days after the last dose of MK-3475 (pembrolizumab). All-cause mortality was tracked from start of treatment through completion of follow-up (up to 5 years after surgery).
Description: The participant not assigned to an arm due to withdrawing before receiving any treatment was not followed for all-cause mortality, serious adverse events, or adverse events.
Arm/Group | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 | Cohort 2: Neoadjuvant MK-3475
All-Cause Mortality (participants affected / at risk) | 14/36 | 2/30
Serious Adverse Events (participants affected / at risk) | 3/36 | 1/30
Other Adverse Events (participants affected / at risk) | 36/36 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 (N=36) | Cohort 2: Neoadjuvant MK-3475 (N=30)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Immune-related hepatitis (Immune system disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Pneumonitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Neoadjuvant MK-3475 and Adjuvant MK-3475 (N=36) | Cohort 2: Neoadjuvant MK-3475 (N=30)
Anemia (Blood and lymphatic system disorders) | 36 | 20
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 4
Cardiac arrest (Cardiac disorders) | 1 | 0
Heart murmur (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 2
Sinus tachycardia (Cardiac disorders) | 10 | 6
Ear pain (Ear and labyrinth disorders) | 5 | 7
Hearing impaired (Ear and labyrinth disorders) | 6 | 3
Left ear fullness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hypoparathyroidism (Endocrine disorders) | 3 | 0
Hypothyroidism (Endocrine disorders) | 9 | 6
Blepharitis (Eye disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Conjuctivitis (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 9 | 3
Diarrhea (Gastrointestinal disorders) | 11 | 3
Dry mouth (Gastrointestinal disorders) | 12 | 1
Dysgeusia (Gastrointestinal disorders) | 8 | 0
Dysphagia (Gastrointestinal disorders) | 20 | 13
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 5
Hemorrhoids (Gastrointestinal disorders) | 0 | 3
Mucositis oral (Gastrointestinal disorders) | 18 | 0
Nausea (Gastrointestinal disorders) | 17 | 4
Odynophagia (Gastrointestinal disorders) | 6 | 2
Oral cavity fistula (Gastrointestinal disorders) | 4 | 2
Oral hemorrhage (Gastrointestinal disorders) | 3 | 1
Oral pain (Gastrointestinal disorders) | 8 | 4
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 2
Chills (General disorders) | 5 | 1
Edema face (General disorders) | 5 | 3
Edema limbs (General disorders) | 9 | 5
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 18 | 7
Fever (General disorders) | 8 | 2
Infusion related reaction (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Malaise (General disorders) | 7 | 0
Neck edema (General disorders) | 7 | 6
Non-cardiac chest pain (General disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Bone infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 4 | 1
Thrush (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 3 | 3
Fall (Injury, poisoning and procedural complications) | 5 | 0
Pain from surgical resection (Injury, poisoning and procedural complications) | 6 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 3
Activated partial thromboplastin time prolonged (Investigations) | 10 | 0
Alanine aminotransferase increased (Investigations) | 6 | 5
Alkaline phosphatase increased (Investigations) | 8 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 7
Blood bilirubin increased (Investigations) | 1 | 1
CPK increased (Investigations) | 1 | 0
Cardiac troponin I increased (Investigations) | 4 | 1
Cholesterol high (Investigations) | 2 | 3
Creatinine increased (Investigations) | 6 | 4
INR increased (Investigations) | 12 | 4
Lymphocyte count decreased (Investigations) | 31 | 11
Neutrophil count decreased (Investigations) | 16 | 2
Platelet count decreased (Investigations) | 13 | 7
Weight loss (Investigations) | 21 | 1
White blood cell count decreased (Investigations) | 20 | 2
Acidosis (Metabolism and nutrition disorders) | 8 | 11
Anorexia (Metabolism and nutrition disorders) | 10 | 2
Dehydration (Metabolism and nutrition disorders) | 8 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 2 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 8 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 21 | 5
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatremia (Metabolism and nutrition disorders) | 11 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 27 | 15
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 15 | 9
Hypomagenesemia (Metabolism and nutrition disorders) | 7 | 2
Hyponatremia (Metabolism and nutrition disorders) | 26 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 14 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness left sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis: upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 9 | 3
Tumor flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 13
Dizziness (Nervous system disorders) | 5 | 1
Dysarthria (Nervous system disorders) | 9 | 6
Dysgeusia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 3
Movements involuntary (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 2
Seizure (Nervous system disorders) | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 1
Tremor (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 9 | 6
Confusion (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 0 | 6
Psychosis (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 7 | 2
Proteinuria (Renal and urinary disorders) | 9 | 3
Renal stones (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 13 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 14 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 | 0
Carotid artery stenosis (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 5 | 1
Hypertension (Vascular disorders) | 30 | 21
Hypotension (Vascular disorders) | 8 | 3
Lymphedema (Vascular disorders) | 12 | 1
Peripheral ischemia (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
After enrollment of 20 patients, an interim analysis was performed to assess the feasibility to achieve the primary endpoint. The trial was amended to: a) close enrollment to cohort 1 b) addition of pTR-2 after neoadjuvant pembrolizumab in all patients as a co-primary endpoint, and c) addition of cohort 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02296684/Prot_SAP_001.pdf